CLINICAL TRIAL: NCT02902926
Title: Comparison of Microbiota and Quality of Life for a Low FODMAPs Versus Standard Dietary Advice in Patients With Irritable Bowel Syndrome
Brief Title: Comparison of Microbiota and Quality of Life for a Low FODMAPs and Standard Dietary in Irritable Bowel Syndrome Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jinsong Wang (Other)
Responsible Party: Sponsor-Investigator, Jinsong Wang, Director of Center for Clincal Epidemiology, Yangzhou University
Organization: Yangzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20160805
Record Dates: First submitted 2016-08-15; First posted 2016-09-16 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Food Habits
MeSH Terms: conditions — Feeding Behavior | interventions — FODMAP Diet

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low FODMAPs Diet (Experimental): 1. Instructed to low FODMAPs diet when patients signed the informed consent.
  2. Answer doubts and correct unhealthy dietary behaviors,such as excessive diet, eating raw, spirits and other excitant food.
  Interventions: Behavioral: Low FODMAPs Diet; Behavioral: Diet instruction
- Diet Instruction (Placebo Comparator): 1.Answer doubts and correct unhealthy dietary behaviors,such as excessive diet, eating raw, spirits and other excitant food.
  Interventions: Behavioral: Diet instruction

INTERVENTIONS:
Behavioral: Low FODMAPs Diet — Instruct to design and eat Low Fermentable，Oligo-，Di-，Mono-saccharides And Polyols(FODMAPs) Diet
  Arms: Low FODMAPs Diet
Behavioral: Diet instruction — Answer the doubt and help the patient get the diet knowlege about the IBS.

SUMMARY:
IBS is a global disease, patients often because of long-term symptoms of recurrent, not timely diagnosis and treatment effect is not ideal and frequent treatment, seriously affect the quality of life, and cause the corresponding economic and social burden.At present，a number of studies suggest that fermentable oligosaccharides, disaccharides and monosaccharides and polyols (FODMAPs) can induce IBS symptoms.Data from large randomized controlled trials are limited, leaving clinicians with the challenge of providing patients with reliable guidance based on minimal evidence.

DETAILED DESCRIPTION:
IBS is a global disease, patients often because of long-term symptoms of recurrent, not timely diagnosis and treatment effect is not ideal and frequent treatment, seriously affect the quality of life, and cause the corresponding economic and social burden.At present，a number of studies suggest that fermentable oligosaccharides, disaccharides and monosaccharides and polyols (FODMAPs) can induce IBS symptoms.Data from large randomized controlled trials are limited, leaving clinicians with the challenge of providing patients with reliable guidance based on minimal evidence.

This study will compare the effect of low FODMAPs diet and usual diet instruction on Intestinal flora, intestinal short chain fatty acids and quality of life by two groups.The results will answer the effect and long-term safety of Low FODMAPs diet.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic criteria for Rome Ⅲ
* IBS patients with diarrhea type
* By endoscopy, X-ray, B ultrasound and laboratory examination to exclude organic disease
* Patients be able to communicate well with the researchers and be willing to participate in the study

Exclusion Criteria:

* Stomach, small intestine, colon surgery history
* irritable bowel disease (IBD) active period, celiac disease
* Alcoholics or drug abuse
* Pregnant or lactating women
* Recent drug users who use defecation
* Have a special diet

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-09; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Microbiota / Short chain fatty acids | Change from baseline Microbiota / Short chain fatty acids at 4 weeks
  The fecal samples of IBS patients were analyzed.

SECONDARY OUTCOMES:
Irritable bowel syndrome severity scoring system scale | Baseline,1,and 3 month post randomization
  Irritable bowel syndrome severity scoring system scale is an integral system for monitoring the severity of IBS in patients with disease severity.The scale is mainly from the degree of abdominal pain, abdominal pain frequency, abdominal distension, defecation satisfaction and the impact of life, according to the 10cm visual scoring method
The Short Form 36 (SF-36) scale | Baseline,1,and 3 month post randomization
  SF-36 is a general scale, at present, the most commonly used evaluation of IBS. It includes 36 items, a total of 8 dimensions
Irritable bowel syndrome quality of life (IBS-QOL) scale | Baseline,1,and 3 month post randomization
  Irritable bowel syndrome quality of life (IBS-QOL) scale is a more extensive application of the specific scale of IBS.
Satisfaction questionnaire | 1,and 3 month post randomization
  To understand the patient's satisfaction with symptom control and diet guidance. The questionnaire included 3 items

CONTACTS AND LOCATIONS:
Overall Officials: Hongcan Shi, Ph.D.,M.D., Study Chair — Medical College
Locations (1):
- YangzhouUniversity, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Canavan C, West J, Card T. Review article: the economic impact of the irritable bowel syndrome. Aliment Pharmacol Ther. 2014 Nov;40(9):1023-34. doi: 10.1111/apt.12938. Epub 2014 Sep 9. PMID 25199904
- [Result] Lovell RM, Ford AC. Global prevalence of and risk factors for irritable bowel syndrome: a meta-analysis. Clin Gastroenterol Hepatol. 2012 Jul;10(7):712-721.e4. doi: 10.1016/j.cgh.2012.02.029. Epub 2012 Mar 15. PMID 22426087
- [Result] Eswaran S, Tack J, Chey WD. Food: the forgotten factor in the irritable bowel syndrome. Gastroenterol Clin North Am. 2011 Mar;40(1):141-62. doi: 10.1016/j.gtc.2010.12.012. PMID 21333905
- [Result] Bohn L, Storsrud S, Tornblom H, Bengtsson U, Simren M. Self-reported food-related gastrointestinal symptoms in IBS are common and associated with more severe symptoms and reduced quality of life. Am J Gastroenterol. 2013 May;108(5):634-41. doi: 10.1038/ajg.2013.105. PMID 23644955
- [Result] Iacovou M, Tan V, Muir JG, Gibson PR. The Low FODMAP Diet and Its Application in East and Southeast Asia. J Neurogastroenterol Motil. 2015 Oct 1;21(4):459-70. doi: 10.5056/jnm15111. PMID 26350937
- [Result] De Giorgio R, Volta U, Gibson PR. Sensitivity to wheat, gluten and FODMAPs in IBS: facts or fiction? Gut. 2016 Jan;65(1):169-78. doi: 10.1136/gutjnl-2015-309757. Epub 2015 Jun 15. PMID 26078292
- [Result] Gibson PR, Varney J, Malakar S, Muir JG. Food components and irritable bowel syndrome. Gastroenterology. 2015 May;148(6):1158-74.e4. doi: 10.1053/j.gastro.2015.02.005. Epub 2015 Feb 11. PMID 25680668
- [Result] Hyland NP, Quigley EM, Brint E. Microbiota-host interactions in irritable bowel syndrome: epithelial barrier, immune regulation and brain-gut interactions. World J Gastroenterol. 2014 Jul 21;20(27):8859-66. doi: 10.3748/wjg.v20.i27.8859. PMID 25083059
- [Result] Jain I, Kumar V, Satyanarayana T. Xylooligosaccharides: an economical prebiotic from agroresidues and their health benefits. Indian J Exp Biol. 2015 Mar;53(3):131-42. PMID 25872243
- [Result] Halmos EP, Power VA, Shepherd SJ, Gibson PR, Muir JG. A diet low in FODMAPs reduces symptoms of irritable bowel syndrome. Gastroenterology. 2014 Jan;146(1):67-75.e5. doi: 10.1053/j.gastro.2013.09.046. Epub 2013 Sep 25. PMID 24076059
- [Result] Bohn L, Storsrud S, Liljebo T, Collin L, Lindfors P, Tornblom H, Simren M. Diet low in FODMAPs reduces symptoms of irritable bowel syndrome as well as traditional dietary advice: a randomized controlled trial. Gastroenterology. 2015 Nov;149(6):1399-1407.e2. doi: 10.1053/j.gastro.2015.07.054. Epub 2015 Aug 5. PMID 26255043
- [Result] Whigham L, Joyce T, Harper G, Irving PM, Staudacher HM, Whelan K, Lomer MC. Clinical effectiveness and economic costs of group versus one-to-one education for short-chain fermentable carbohydrate restriction (low FODMAP diet) in the management of irritable bowel syndrome. J Hum Nutr Diet. 2015 Dec;28(6):687-96. doi: 10.1111/jhn.12318. Epub 2015 Apr 14. PMID 25871564
- [Result] Marsh A, Eslick EM, Eslick GD. Does a diet low in FODMAPs reduce symptoms associated with functional gastrointestinal disorders? A comprehensive systematic review and meta-analysis. Eur J Nutr. 2016 Apr;55(3):897-906. doi: 10.1007/s00394-015-0922-1. Epub 2015 May 17. PMID 25982757
- [Result] Chumpitazi BP, Cope JL, Hollister EB, Tsai CM, McMeans AR, Luna RA, Versalovic J, Shulman RJ. Randomised clinical trial: gut microbiome biomarkers are associated with clinical response to a low FODMAP diet in children with the irritable bowel syndrome. Aliment Pharmacol Ther. 2015 Aug;42(4):418-27. doi: 10.1111/apt.13286. Epub 2015 Jun 24. PMID 26104013
- See also: Monash University, D.o.G., The Monash University low FODMAP diet app. Melbourne Australia: Central Clinical School 2015 [updated 28 May 2015; cited 2015 4 June]. — http://www.med.monash.edu.au/cecs/gastro/fodmap/iphone-app.html